CLINICAL TRIAL: NCT01699659
Title: The Efficacy and Safety of the United Allergy Service (UAS) Immunotherapy Protocol
Brief Title: The Efficacy & Safety of the UAS Immunotherapy Protocol
Status: Completed | Type: Observational
Sponsor: United Allergy Services (Industry)
Responsible Party: Principal Investigator, Frederick M. Schaffer, MD, Chief Medical Officer, United Allergy Services
Other Study IDs: UAS protocol #1; UAS protocol #1 (Other Grant/Funding Number: United Allergy Services)
Record Dates: First submitted 2012-09-10; First posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Perennial Allergic Rhinitis With Seasonal Variation
Keywords: Allergic Rhinitis; Allergen Immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Desensitization, Immunologic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: allergen immunotherapy — allergy shots
  Other Names: allergy shots

SUMMARY:
Hypothesis: The UAS Immunotherapy protocol is efficacious and at least as efficacious as protocols described in the Allergy literature.

DETAILED DESCRIPTION:
Patients will be assessed for efficacy of the immunotherapy protocol by completing Consented-IRB approved clinical, medication, quality of life survey questions comparing current status while on therapy in contrast to 12 months before the inception of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Allergic rhinitis between 18 and 65 years old who have chosen to undergo immunotherapy.

Exclusion Criteria:

* No beta blocker use,
* no pregnancy,
* no systemic steroids,
* no severe asthma/copd,
* no severe collagen vascular disorders,
* no neoplastic or uncontrolled seizure activity,
* no previous anaphylaxis, no significant cardiovsacular disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with allergic rhinitis pre and post immunotherapy (1 to 2 years).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
change in symptom scores from 12 months before therapy initiation in contrast to determination during 1 to 2 years of therapy (retrospective). | Assessment contrasts current status (at 1 to 2 years of therapy) to a point 12 months prior to the onset of therapy.
  Enrolled patients completed surveys pertinent to symptom scores, contrasting current status on immunotherapy compared (by recall) to a 12 month time point prior to initiation of therapy.

SECONDARY OUTCOMES:
Changes in medication plus symptom aggregate score. | Assessment contrasts current status (at 1 to 2 years of therapy) to a point 12 months prior to the onset of therapy.
  Aggregate Medication and Symptom surveys were compared to determine changes from a 12 month time point prior to inception of therapy to current time point of 1 to 2 years of therapy.

OTHER OUTCOMES:
Quality of Life (QOL) scores | Assessment contrasts current status (at 1 to 2 years of therapy) to a point 12 months prior to the onset of therapy
  QOL scores will be calculated after one to 2 years of therapy and contrasted with QOL reflecting status 12 months prior to initiation of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick M Schaffer, M.D., Principal Investigator — United Allergy Services
Locations (1):
- UAS, San Antonio, Texas, United States